CLINICAL TRIAL: NCT06746077
Title: INSPIRE CHILD: Investigating Novel Strategies in Pediatric Immune Responses and Microbiome Environment: Comprehensive Lung Disease Investigation in Children
Brief Title: Investigating Novel Strategies in Pediatric Immune Responses and Microbiome Environment: Comprehensive Lung Disease Investigation in Children.
Acronym: INSPIRE CHILD
Status: Enrolling by invitation | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Sune Rubak, Consultant, Associate Professor, Aarhus University Hospital
Other Study IDs: VEK j.nr. 1-10-72-8-24
Record Dates: First submitted 2024-09-27; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Lung Diseases
Keywords: Pediatric; Lung Disease; Microbiome; Cytokine; Inflammation; Immune Cell; Bacteria; Asthma; Coughing; Immunophenotype; Bronchiectasis; Bronchoscopy; BAL; Bronchoalveolar lavage; Diffuse Lung Disease; Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases; Inflammation; Asthma; Cough; Bronchiectasis; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage (BAL)-samples will be collected as well as a blood sample.
  Both are kept in storage in a biobank for further research projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The INSPIRE CHILD-study is a clinical research project focused on understanding lung diseases in children. The study aims to explore how the presence of certain bacteria, immune responses, and inflammatory markers in the lungs are connected to different lung diseases in pediatric patients.

Background:

Lung diseases in children can have long-lasting effects on their health, not only during childhood but also as they grow into adults. However, the specific causes and mechanisms behind these diseases are not yet fully understood. The INSPIRE CHILD-study is designed to investigate whether children with various lung conditions have distinct differences in the types of bacteria, immune system activity, and inflammation in their lungs.

Hypothesis:

Different lung diseases in children are hypothesized to be associated with unique patterns of bacteria, immune responses, and inflammation in the lungs By studying these patterns, the investigators hope to gain new insights that could lead to better diagnostic tools and more personalized treatments for children suffering from lung diseases.

Children already scheduled to undergo bronchoscopy are included in the study. A small sample of fluid from the lungs is collected, and the sample is analyzed for bacteria, immune markers, and signs of inflammation. This research could pave the way for improved care and treatment for young patients with lung conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from new-born to 17 years of age.
* Diagnosed with or being assessed for a lung disease.
* Possible to sample at least 2 ml of BAL-fluid besides the scheduled amount during the bronchoscopy.

Exclusion Criteria:

* Age older than 17 years.
* Not undergoing diagnosis at Childrens Center for Pulmonary and Allergic diseases.
* Failure to meet the requirement of being able to sample an additional 2 ml of BAL-fluid.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 200 children/adolescents with lung disease undergo bronchoscopy yearly at Childrens Center for Pulmonary and Allergic diseases, Aarhus University Hospital. All patients are on clinical indication already scheduled for bronchoscopy and BAL. Participants are recruited from this group of patients if they comply with the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytokines | Day 0 (Subsequent to study inclusion)
  Legendplex assay for measuring cytokines in bronchoalveolar lavage fluid and plasma (e.g. IL-1-beta, IL-1RA, IL-2, IL-6, IL-8, IL-10, IL-17, IL-18, IL-33, IL-35, TGF-beta, TNF-alpha)
Immunophenotype | Day 0 (Subsequent to study inclusion)
  Using flow cytometry to investigate immune cells:
  e.g. Neutrophils, Eosinophils, Monocytes, NK-cells, B-cells, CD4+-T-cells, CD8+-T-cells
Lung microbiome | Day 0 (Subsequent to study inclusion)
  We seek to investigate whether it is feasible to map the microbiome, virome and mycobiome of the pediatric lung from BAL-fluid.
  The study will investigate and report findings of bioinformatics analysis.

SECONDARY OUTCOMES:
Concentration range for selected interleukins in BAL-fluid | Day 0 (Subsequent to study inclusion)
Lung disease association | Through study completion, an average of 2 year
  Can we associate a specific profile of findings with a particular pediatric lung disease?
Clinical symptoms | 2 weeks prior to enrollment
  2 weeks prior to date of inclusion/bronchoscopy, the subjects medical history is reviewed for the following:
  Characterization of cough
  Respiratory distress
  Functional limitations (due to respiratory distress) (acc. to age)
  Fever (temperature above 38.0 C)
  Breath sounds
  Urgent need for medication

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Center for Pulmonary and Allergic diseases, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data that underlie the results reported in study articles (text, tables, figures, and appendices).
  The laws related to the handling of personal data will be followed and results are processed in accordance with the General Data Protection Regulation (GDPR) and the Danish Data Protection Act (Databeskyttelsesforordningen and Databeskyttelsesloven).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the study has been finalized.
Access Criteria: Researchers who provide a methodologically sound proposal.